CLINICAL TRIAL: NCT02230670
Title: A Multicenter, Double-Blind, Placebo Controlled Study to Evaluate the Safety, Tolerability and Efficacy of IDN-6556 in Subjects With Liver Cirrhosis
Brief Title: A Study of IDN-6556 in Subjects With Liver Cirrhosis
Acronym: LC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDN-6556-10
Record Dates: First submitted 2014-08-28; First posted 2014-09-03 (Estimated); Results first posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Liver Cirrhosis; Hepatic Cirrhosis
Keywords: Liver Cirrhosis; Hepatic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IDN-6556 (Experimental): 25 mg BID of IDN-6556
  Interventions: Drug: IDN-6556
- Placebo (Placebo Comparator): Placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IDN-6556 — 25 mg BID
  Other Names: emricasan; PF-03491390
  Arms: IDN-6556
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter study to see if treatment with IDN-6556 can help improve the liver function of patients with liver cirrhosis with Model for End-Stage Liver Disease scores between 11-18.

DETAILED DESCRIPTION:
Numerous studies have shown that caspase cleaved cytokeratin 18 (cCK18) is elevated in the serum of liver disease patients and has been associated with disease severity, thus associating both excessive apoptosis and caspase activity with disease. Studies have also shown that caspase cleaved cytokeratin 18 is generally elevated to an even greater degree in cirrhosis than in other liver diseases. In addition, increasing stages of cirrhosis from Child-Pugh A, Child-Pugh B to Child-Pugh C are associated with progressively higher levels of caspase cleaved cytokeratin 18. Therefore, it appears that apoptosis and caspase activity tend to correlate with the stage of cirrhosis. A caspase inhibitor like IDN-6556 could have clinical utility by reducing the rate of apoptosis in cirrhotic patients and potentially reduce the progression of disease as determined by clinical markers of progression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of minimum adult legal age (according to local laws for signing the informed consent document), able to provide written informed consent, and able to understand and willing to comply with the requirements of the study
* Clinical, radiological, or biochemical evidence of liver cirrhosis
* Model for End-Stage Liver Disease (MELD) Score of 11 to 18 during the Screening period
* Willingness to utilize two reliable forms of contraception (for both males and females of childbearing potential) from Screening to one month after the last dose of study drug.

Exclusion Criteria:

* Known infection with human immunodeficiency virus (HIV)
* Auto-immune hepatitis
* Subjects with evidence of uncontrolled infection, defined as persistent bacterial culture positivity despite adequate antibiotic therapy
* HCV infected subjects who are receiving or plan to receive anti-viral therapy during the study
* Untreated esophageal varices with high risk stigmata for hemorrhage
* Variceal hemorrhage within 3 months of Screening
* Ascites not adequately controlled on stable background medication
* Other non-liver organ failure
* Child-Pugh score of 10-15 (Child-Pugh C classification)
* Use of vasoactive drugs (at or within 3 months of Screening) that may impair hepatic blood flow
* Change in dose or regimen within 3 months of Screening of:

  1. Fibrates or statins
  2. Angiotensin II receptor antagonist or angiotensin converting enzyme (ACE) inhibitor
* Use of chronic anticoagulation therapy including but not limited to Vitamin K/Factor Xa antagonists/inhibitors
* Use of the following drugs within 2 months of Screening:

  1. Systemic corticosteroids
  2. Known or suspected use of illicit drugs or drugs of abuse (allowed if medically prescribed or indicated)
* Concomitant pancreatitis
* Active inflammatory bowel disease
* Diagnosed or suspected systemic lupus erythematosus (SLE) and/or rheumatoid arthritis (RA)
* Subjects with active or history of malignancies other than hepatocellular carcinoma (HCC) within Milan criteria or curatively treated skin cancer (basal cell or squamous cell carcinomas), unless adequately treated or in complete remission for five or more years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Hagerty, MD, Study Chair — Conatus Pharmaceuticals Inc.
Locations (28):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Scripps Clinic, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Cedar-Sinai Medical Center, Los Angeles, California
  - Univeristy of California, San Diego, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Cente, Maywood, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Henry Ford Hospital, Detroit, Michigan
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - NYU Medical Center, New York, New York
  - Mt. Sinai School of Medicine, New York, New York
  - University of Cincinnati Physicians Company, LLC, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - UT Health Science Center at Houston, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Bon Secours Mary Immaculate Hospital, Newport News, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Inc., Richmond, Virginia

REFERENCES:
- [Derived] Frenette CT, Morelli G, Shiffman ML, Frederick RT, Rubin RA, Fallon MB, Cheng JT, Cave M, Khaderi SA, Massoud O, Pyrsopoulos N, Park JS, Robinson JM, Yamashita M, Spada AP, Chan JL, Hagerty DT. Emricasan Improves Liver Function in Patients With Cirrhosis and High Model for End-Stage Liver Disease Scores Compared With Placebo. Clin Gastroenterol Hepatol. 2019 Mar;17(4):774-783.e4. doi: 10.1016/j.cgh.2018.06.012. Epub 2018 Jun 18. PMID 29913280

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 140 subjects from 26 US sites were screened, of whom 87 subjects were randomized. One subject randomized to placebo withdrew from the study before taking study drug. Disposition data is provided for the initial 3-month randomized, placebo-controlled phase on which the primary efficacy and safety analyses were based
Groups:
- Placebo: Placebo BID
  Placebo
Period: Overall Study
Arm/Group | IDN-6556 | Placebo
Started | 44 | 42 (One subject randomized to placebo withdrew from the study before receiving any study treatment.)
Completed | 40 | 34
Not Completed | 4 | 8
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Progression to Child-Pugh C | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDN-6556 | Placebo | Total
Number analyzed (Participants) | 44 | 42 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 34 | 69
  >=65 years | 9 | 8 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 32
  Male | 24 | 30 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 11 | 17
  Not Hispanic or Latino | 38 | 30 | 68
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 39 | 37 | 76
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Month 3 in cCK18/M30
Description: Baseline, Month 3, and change between for cCK18/M30
Time Frame: 3 months
Population: FAS
Measure: Median (Full Range); unit: U/L
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 44 | 42
U/L
  Baseline | 293.5 [66 to 1857] | 257.5 [104 to 6994]
  Month 3 | 288.5 [39 to 1583] | 285.0 [115 to 19710]

2. Primary Outcome: Change From Baseline at Month 3 in cCK18/M30
Description: Data was log-transformed for analysis purposes
Time Frame: 3 months
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 44 | 42
U/L
  Log-transformed Values | -0.049 (0.057) | 0.090 (0.058)
  Percent (%) Relative Change | -4.6 (5.9) | 9.3 (5.9)
Statistical Analysis 1: Comparison: IDN-6556 vs Placebo; Analysis was conducted using an ANCOVA model adjusting for baseline value; Test type: Superiority; p = 0.091, ANCOVA; Mean Difference (Final Values) = -0.140, 95% CI 2-sided [-0.302 to 0.023], Standard Error of Mean 0.0817
Statistical Analysis 2: Comparison: IDN-6556 vs Placebo; The analysis was conducted using an ANCOVA model adjusting for baseline value, baseline MELD score, and etiology. The significance was assessed using Type II Sums of Squares from this ANCOVA model; Test type: Superiority; p = 0.041, ANCOVA; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.41 to 0.01], Standard Error of Mean .210

3. Secondary Outcome: Change From Baseline to Month 3 in MELD Score
Description: The Model for End-Stage Liver Disease (MELD) is a scoring system for assessing the severity of chronic liver disease and uses the subject's values for total bilirubin, serum creatinine, and the international normalized ratio (INR) for prothrombin time to predict survival. MELD is calculated according to the following formula:
  MELD = 3.78×ln[serum bilirubin (mg/dL)] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43
  MELD scores are reported as whole numbers, so the result of the equation above is rounded. Notes: If the patient has been dialyzed twice within the last 7 days, then the value for serum creatinine used should be 4.0. Any value less than one is given a value of 1 (i.e. if bilirubin is 0.8, a value of 1.0 is used) to prevent the occurrence of scores below 0 (the natural logarithm of 1 is 0, and any value below 1 would yield a negative result). The higher the MELD score the more severe the disease state.
Time Frame: 3 Months
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 44 | 42
units on a scale | -0.10 (0.234) | 0.15 (0.239)
Statistical Analysis 1: Comparison: IDN-6556 vs Placebo; Analysis was conducted using an ANCOVA model adjusting for baseline value; Test type: Superiority; p = 0.466, ANCOVA; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.91 to 0.42], Standard Error of Mean 0.333
Statistical Analysis 2: Comparison: IDN-6556 vs Placebo; BL MELD >= 15 subgroup results (N=19), as analyzed from the adjusted analysis ANCOVA model adjusting for baseline value, baseline MELD score, and etiology; Test type: Superiority; p = 0.003, ANCOVA; calculated from the estimated least square means for the treatment by BL MELD category interaction term; Median Difference (Final Values) = -2.19, 95% CI 2-sided [-3.61 to -0.77], Standard Error of Mean 1.42
Statistical Analysis 3: Comparison: IDN-6556 vs Placebo; NASH Etiology subgroup results (N=20), as analyzed from the adjusted analysis ANCOVA model adjusting for baseline value, baseline MELD score, and etiology; Test type: Superiority; p = 0.029, ANCOVA; calculated from the estimated least square means for the treatment by etiology interaction term; Median Difference (Final Values) = -1.6, 95% CI 2-sided [-3.09 to -0.17], Standard Error of Mean 1.46

ADVERSE EVENTS:
Time Frame: Adverse events were collected in a blinded fashion from baseline to Month 3. Double-blind adverse events are presented here
Groups:
- IDN-6556 (Baseline-Month 3): 25 mg BID of IDN-6556 (Baseline-Month 3).
- Placebo (Baseline-Month 3): Placebo BID (Baseline-Month 3)
Arm/Group | IDN-6556 (Baseline-Month 3) | Placebo (Baseline-Month 3)
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/42
Serious Adverse Events (participants affected / at risk) | 6/44 | 5/42
Other Adverse Events (participants affected / at risk) | 34/44 | 30/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDN-6556 (Baseline-Month 3) (N=44) | Placebo (Baseline-Month 3) (N=42)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Peritontis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Accidential overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site heamorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Convulsions (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary alveolar haemorrage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDN-6556 (Baseline-Month 3) (N=44) | Placebo (Baseline-Month 3) (N=42)
abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3)
arthralgia (General disorders) | 3 (3) | 0 (0)
ascites (Gastrointestinal disorders) | 1 (2) | 3 (3)
fatigue (Metabolism and nutrition disorders) | 4 (4) | 6 (7)
headache (Nervous system disorders) | 7 (8) | 3 (4)
hepatic encephalopathy (Nervous system disorders) | 5 (7) | 2 (3)
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
nausea (Gastrointestinal disorders) | 7 (8) | 4 (5)
oedema peripheral (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
vomiting (Gastrointestinal disorders) | 5 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less